CLINICAL TRIAL: NCT00316251
Title: Application of Specific Frequencies to Stimulate the Spinocerebellar Tract in Subjects With Unilateral Dysafferentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR0403060006
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-04

CONDITIONS: Somatosensory Disorders
Keywords: Somatosensory dysfunction
MeSH Terms: conditions — Somatosensory Disorders

INTERVENTIONS:
Device: Vibration Plate Therapy

SUMMARY:
The purpose of this study is to determine the effects of Power Plate vibration therapy on balance as measured by the NeuroCom Balance Master.

DETAILED DESCRIPTION:
Acute and chronic equilibrium disorders result in over five million patient visits per year in the United States with unknown additional individuals not seeking care. Symptoms of dizziness, vertigo, and lack of balance are among the most common symptoms reported to physicians. Equilibrium disorders not exclusively due to visual or vestibular conditions are typically due to problems in proprioception. Proprioception is the specialized sensory modality that informs the body as to movement, position, and spatial orientation through mechanisms that track sensations accompanying joint movement and position. Mechanoreceptors in joints, along with vestibular, visual, muscle spindle, Golgi tendon organ, ligament and tendon sensory receptors, comprise the propriosensory system, which conveys information to the motor system to maintain equilibrium on a reflexive, automatic basis. Alterations in somatosensory input from mechanoreceptors have been identified as causing aberrant muscle firing patterns.

The NeuroCom Balance Master is an FDA approved device designed to both measure and treat balance problems and evaluate the neuromuscular control by quantifying the ability to maintain dynamic postural stability. The NeuroCom Unit is a microprocessor controlled balance unit that provides quantitative data regarding the patient's ability to control the platform. This unit is widely used throughout the country in both university and clinical settings to help patients restore their balance.

ELIGIBILITY:
Inclusion Criteria:

* Logan student, staff, or faculty with no history of ankle injury
* Ages 18 - 60 years old
* Logan student, staff, or faculty with no history of ankle surgery
* No visual or vestibular condition that would affect balance

Exclusion Criteria:

* Systemic illnesses that have an adverse effect on balance
* Local infection, injury, or other malignancy affecting the lower extremity
* Any unstable joints of the lower extremity
* Any spinal manipulation within 48 hours
* Prescription or herbal muscle stimulants, relaxants, etc. that could affect balance
* Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2
Dates: Start 2006-04; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Enix, DC, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States